CLINICAL TRIAL: NCT00662818
Title: A Multicenter, Randomized, Double-Blind, Placebo- and Active Controlled, Crossover Study to Evaluate the Safety and Efficacy of MK-0974 in the Treatment of Acute Migraine in Patients With Stable Vascular Disease
Brief Title: Telcagepant (MK-0974) Treatment of Migraine in Participants With Stable Vascular Disease (MK-0974-034)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0974-034; MK-0974-034 (Other: Merck Protocol Number); 2007_545 (Other: Telerx ID Number)
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-09

CONDITIONS: Migraine Disorders; Heart Disease; Cerebrovascular Accident; TIA (Transient Ischemic Attack); Vascular Diseases; Peripheral Vascular Diseases
MeSH Terms: conditions — Migraine Disorders; Heart Diseases; Stroke; Ischemic Attack, Transient; Vascular Diseases; Peripheral Vascular Diseases | interventions — telcagepant; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telcagepant 300 mg→Acetaminophen/Paracetamol 1000 mg (Experimental): Participants receive up to 12 doses of telcagepant (280 mg tablet/capsule 300 mg), orally, and placebo to acetaminophen/paracetamol (APAP) (2- 500 mg dry filled capsules), orally, for up to 12 migraine attacks in Period 1 (6 weeks). Participants receive APAP and placebo to telcagepant for up to 12 doses, for up to 12 migraine attacks in Period 2 (6 weeks). The participant may take a blinded optional second dose of study medication or their own rescue medication if 2 hours after initial treatment, the participant still has a moderate or severe migraine headache or if the headache has returned.
  Interventions: Drug: Telcagepant; Drug: Acetaminophen/Paracetamol; Drug: Placebo to Telcagepant; Drug: Placebo to Acetaminophen/Paracetamol
- Placebo and APAP 1000 mg→Telcagepant 300 mg (Experimental): Participants receive 1 dose of placebo to APAP and placebo to telcagepant for the first migraine attack and then up to 11 doses of APAP and placebo to telcagepant for up to 11 migraine attacks in Period 1 (6 weeks). Participants receive up to 12 doses of telcagepant and placebo to APAP for up to 12 migraine attacks in Period 2 (6 weeks). The participant may take a blinded optional second dose of study medication or their own rescue medication if 2 hours after initial treatment, the participant still has a moderate or severe migraine headache or if the headache has returned.
  Interventions: Drug: Telcagepant; Drug: Acetaminophen/Paracetamol; Drug: Placebo to Telcagepant; Drug: Placebo to Acetaminophen/Paracetamol

INTERVENTIONS:
Drug: Telcagepant — Telcagepant (MK-0974) (300 mg soft gel capsules or 280 mg tablets)
Drug: Acetaminophen/Paracetamol — Acetaminophen/Paracetamol (500 mg X 2 dosage units)
Drug: Placebo to Telcagepant — Placebo 300 mg soft gel capsules or placebo 280 mg tablet.
Drug: Placebo to Acetaminophen/Paracetamol — Placebo to acetaminophen/paracetamol (500 mg X 2 dosage units)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of telcagepant in the treatment of acute migraine in participants with stable vascular disease. Acetaminophen/paracetamol (APAP) will be used as an active comparator in this study. The primary hypothesis of this study is that telcagepant 300 mg is superior to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary artery disease for 3 months or more
* 18 years of age or older with a history of migraine with or without aura
* Must use acceptable contraception throughout the study

Exclusion Criteria:

* Pregnant, breast-feeding, or planning to become pregnant during this study
* 50 years of age or older when migraines began
* Other pain syndromes that might interfere with study assessments, uncontrolled psychiatric conditions, dementia, or significant neurological disorders (other than migraine)
* History of gastric, or small intestinal surgery, or has a disease that causes malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-03-17 (Actual); Primary Completion 2009-09-02 (Actual); Study Completion 2009-09-02 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Ho TW, Ho AP, Chaitman BR, Johnson C, Mathew NT, Kost J, Fan X, Aurora SK, Brandes JL, Fei K, Beebe L, Lines C, Krucoff MW. Randomized, controlled study of telcagepant in patients with migraine and coronary artery disease. Headache. 2012 Feb;52(2):224-35. doi: 10.1111/j.1526-4610.2011.02052.x. Epub 2012 Jan 6. PMID 22221076
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-034&kw=0974-034&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Telcagepant 300 mg→Acetaminophen/Paracetamol 1000 mg: Participants receive up to 12 doses of telcagepant (300 mg capsule/280 mg tablet), orally, and placebo to acetaminophen/paracetamol (APAP) (2- 500 mg dry filled capsules), orally, for up to 12 migraine attacks in Period 1 (6 weeks). Participants receive APAP and placebo to telcagepant for up to 12 doses, for up to 12 migraine attacks in Period 2 (6 weeks).
- Placebo and APAP 1000 mg→Telcagepant 300 mg: Participants receive 1 dose of placebo to APAP and placebo to telcagepant for the first migraine attack and then up to 11 doses of APAP and placebo to telcagepant for up to 11 migraine attacks in Period 1 (6 weeks). Participants receive up to 12 doses of telcagepant and placebo to APAP for up to 12 migraine attacks in Period 2 (6 weeks).
Period: Period 1 (6 Weeks)
Arm/Group | Telcagepant 300 mg→Acetaminophen/Paracetamol 1000 mg | Placebo and APAP 1000 mg→Telcagepant 300 mg
Started | 84 | 81
Treated | 56 | 58
Completed | 56 | 58
Not Completed | 28 | 23
Period: Wash-Out (14 Days)
Arm/Group | Telcagepant 300 mg→Acetaminophen/Paracetamol 1000 mg | Placebo and APAP 1000 mg→Telcagepant 300 mg
Started | 56 | 58
Completed | 51 | 53
Not Completed | 5 | 5
Period: Period 2 (6 Weeks)
Arm/Group | Telcagepant 300 mg→Acetaminophen/Paracetamol 1000 mg | Placebo and APAP 1000 mg→Telcagepant 300 mg
Started | 51 | 53
Completed | 38 | 41
Not Completed | 13 | 12

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Telcagepant 300 mg→APAP 1000 mg: Participants receive up to 12 doses of telcagepant (280 mg tablet/capsule 300 mg), orally, and placebo to acetaminophen/paracetamol (APAP) (2- 500 mg dry filled capsules), orally, for up to 12 migraine attacks in Period 1 (6 weeks). Participants receive APAP and placebo to telcagepant for up to 12 doses, for up to 12 migraine attacks in Period 2 (6 weeks).
- Total: Total of all reporting groups
Arm/Group | Telcagepant 300 mg→APAP 1000 mg | Placebo and APAP 1000 mg→Telcagepant 300 mg | Total
Number analyzed (Participants) | 56 | 58 | 114
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (10.1) | 55.7 (10.0) | 56.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pain Freedom at 2 Hours Post-dose (Period 1, Migraine Attack 1)
Description: Pain Freedom (PF) at 2 hours post-dose (Period 1, Attack 1) defined as a decrease from a moderate or severe migraine headache (Grade 2 or 3) at baseline to no pain (Grade 0). Headache severity was subjectively rated by the participant at predefined time points on a scale of Grade 0 to Grade 3: Grade 0 - No pain; Grade 1 - Mild pain; Grade 2 - Moderate Pain; and Grade 3 - Severe Pain.
Time Frame: 2 hours post-dose (Up to 6 weeks)
Population: The full-analysis set (FAS) included participants treated for a migraine attack. Participants had both a baseline value and at least 1 post-dose efficacy measurement for pain severity prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline pain score or post-dose data through 2 hours.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Telcagepant 300 mg: Participants receiving telcagepant
- Placebo: Participants receiving placebo
Arm/Group | Telcagepant 300 mg | Placebo
Number analyzed (Participants) | 52 | 53
Percentage of participants | 25.0 [14.0 to 38.9] | 18.9 [9.4 to 32.0]
Statistical Analysis 1: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p = 0.329, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.62 to 4.25]

2. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Post-dose (Period 1, Migraine Attack 1)
Description: Pain Relief (PR) at 2 hours post-dose (first migraine attack), with pain relief defined as a reduction in headache severity from Grade 3/2 at baseline to Grade 1/0 at 2 hours post-dose. Headache severity was subjectively rated by the participant at predefined time points on a scale of Grade 0 to Grade 3: Grade 0 - No pain; Grade 1 - Mild pain; Grade 2 - Moderate Pain; and Grade 3 - Severe Pain.
Time Frame: 2 hours post-dose (Up to 6 weeks)
Population: The FAS Population included participants treated that migraine attack, and had both a baseline value and at least 1 post-dose efficacy measurement for pain severity prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline pain score or post-dose data through 2 hours.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Telcagepant 300 mg | Placebo
Number analyzed (Participants) | 52 | 53
Percentage of Participants | 63.5 [49.0 to 76.4] | 56.6 [42.3 to 70.2]
Statistical Analysis 1: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p = 0.420, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.59 to 3.50]

3. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE) Within 14 Days Post-dose
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Within 14 days of any dose of study medication (Up to 16 weeks)
Population: All-Patients-as-Treated (APaT) population consisted of all participants who received at least 1 dose of study medication were included in the treatment group according to the medication actually received.
Measure: Number; unit: Participants
Groups:
- Acetaminophen/Paracetamol (APAP): Participants receiving APAP
Arm/Group | Telcagepant 300 mg | Acetaminophen/Paracetamol (APAP)
Number analyzed (Participants) | 98 | 86
Participants | 21 | 14

4. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an AE Within 48 Hours Post-dose
Description: as for outcome 3
Time Frame: Up to 48 hours post-dose (Up to 14 weeks)
Population: The APaT Population consisted of all participants who received at least 1 dose of study medication were included in the treatment group according to the medication actually received.
Measure: Number; unit: Participants
Groups:
- APAP: Participants receiving APAP
Arm/Group | Telcagepant 300 mg | APAP
Number analyzed (Participants) | 98 | 86
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With a Confirmed Vascular Event Within 48 Hours Post-dose
Description: Confirmed Vascular Event included cardiac events, cerebrovascular events, and peripheral vascular events.
Time Frame: Up to 48 hours after the dose of any study medication (Up to 14 weeks)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Telcagepant 300 mg | APAP
Number analyzed (Participants) | 98 | 86
Participants | 0 | 0

6. Secondary Outcome: Percentage of Participants With Absence of Phonophobia at 2 Hours Post-dose (Period 1, Migraine Attack 1)
Description: The participant recorded whether phonophobia (sensitivity to sound) was present or absent at each of the predefined time points.
Time Frame: 2 hours post-dose (Up to 6 weeks)
Population: The FAS population included participants treated that migraine attack, and had both a baseline value and at least 1 post-dose efficacy measurement for phonophobia prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline phonophobia score or post-dose data through 2 hours.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Telcagepant 300 mg | Placebo
Number analyzed (Participants) | 52 | 53
Percentage of participants | 65.4 [50.9 to 78.0] | 58.5 [44.1 to 71.9]
Statistical Analysis 1: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p = 0.648, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.52 to 2.85]

7. Secondary Outcome: Percentage of Participants With Absence of Photophobia at 2 Hours Post-dose (Period 1, Migraine Attack 1)
Description: The participant recorded whether photophobia (sensitivity to light) was present or absent at each of the predefined time points.
Time Frame: 2 Hours post-dose (Up to 6 weeks)
Population: The FAS population included participants treated that migraine attack, and had both a baseline value and at least 1 post-dose efficacy measurement for photophobia prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline photophobia score or post-dose data through 2 hours.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Telcagepant 300 mg | Placebo
Number analyzed (Participants) | 52 | 53
Percentage of Participants | 53.8 [39.5 to 67.8] | 58.5 [44.1 to 71.9]
Statistical Analysis 1: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p = 0.647, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.31 to 2.07]

8. Secondary Outcome: Percentage of Participants With Absence of Nausea at 2 Hours Post-dose (Period 1, Migraine Attack 1)
Description: The participant recorded whether nausea was present or absent at each of the predefined time points.
Time Frame: 2 hours post-dose (Up to 6 weeks)
Population: The FAS population included participants treated that migraine attack, and had both a baseline value and at least 1 post-dose efficacy measurement for nausea prior to, or including, the 2-hour time point. Participants were excluded from this analysis who did not have a baseline nausea score or post-dose data through 2 hours.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Telcagepant 300 mg | Placebo
Number analyzed (Participants) | 52 | 53
Percentage of Participants | 80.8 [67.5 to 90.4] | 69.8 [55.7 to 81.7]
Statistical Analysis 1: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p = 0.201, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.73 to 4.60]

9. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom (SPF) at 2 to 24 Hours Post-dose
Description: SPF from 2 to 24 hours post-dose is defined as PF at 2 hours, with no administration of either rescue medication or the optional second dose and with no occurrence thereafter of a mild/moderate/severe headache during the 2 to 24 hours after dosing with the study medication.
Time Frame: Up to 24 hours post-dose (Up to 14 weeks)
Population: The FAS population was participants treated that migraine attack, and had both a baseline value and at least 1 post-dose efficacy measurement for pain severity prior to, or including, the 2-hr. time point. Participants were excluded from this analysis for not having a baseline pain score, post-dose data through 24 hrs, or a recurrence question.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Telcagepant 300 mg | Placebo
Number analyzed (Participants) | 52 | 52
Percentage of Participants | 19.2 [9.6 to 32.5] | 15.4 [6.9 to 28.1]
Statistical Analysis 1: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p = 0.579, Regression, Logistic; Computed using a logistic regression model adjusting for geographic region, baseline migraine severity, and age; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.47 to 3.85]

ADVERSE EVENTS:
Time Frame: Up to 48 hours post-dose (Up to 14 weeks)
Groups:
- Telcagepant: Participants receiving telcagepant
- Acetaminophen/Paracetamol: Participants receiving acetaminophen/paracetamol
Arm/Group | Telcagepant | Acetaminophen/Paracetamol
Serious Adverse Events (participants affected / at risk) | 1/98 | 0/86
Other Adverse Events (participants affected / at risk) | 0/98 | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telcagepant (N=98) | Acetaminophen/Paracetamol (N=86)
Psychotic disorder (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.